CLINICAL TRIAL: NCT02107469
Title: A Randomized Placebo-compared Study on Efficiency of Two Different Administration Forms of Phyllanthus Niruri and Sida Cordifolia in Patients With Diabetic Peripheral Polyneuropathy
Brief Title: A Study of Phyllanthus Niruri and Sida Cordifolia in Diabetic Peripheral Polyneuropathy
Acronym: VEDICINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosenberg European Academy of Ayurveda (Other)
Collaborators: EUROPEAN PROFESSIONAL ASSOCIATION OF AYURVEDA PRACTITIONERS AND THERAPISTS (Unknown)
Responsible Party: Principal Investigator, Prof. S.N. Gupta, Superintendent of P.D. Patel Ayurveda Hospital Nadiad, Gujarat, India, Rosenberg European Academy of Ayurveda
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NADIAD 2014
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Diabetic Polyneuropathy; Diabetic Neuralgia; Diabetic Neuropathies; Diabetic Neuropathy
Keywords: Diabetic Polyneuropathy; Diabetic; Polyneuropathy; Ayurvedic; Ayurveda; Neuralgia; Diabetic Neuralgia; Sida cordifolia; Phyllanthus Niruri; Phyllanthus Amarus; Extracts; Extract; Crude Herb; Crude; Herb; Herbal; Herbal Extract; Decoction; Churna; Powder; Bala; Bhumyamalaki; Tamalaki
MeSH Terms: conditions — Diabetic Neuropathies; Polyneuropathies; Neuralgia | interventions — 4-bromobenzoyl-(alpha-aminoisobutyric acid)(5)-leucyl-(alpha-aminoisobutyric acid)(2)-methoxy; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ancient herbal treatment (Experimental): Phyllanthus niruri 3g fine dry powder 3 times a day with warm water before meals for 8 weeks
  Sida cordifolia 7g coarse dry powder 2 times a day prepared as traditional decoction before meals for 8 weeks. Decoction: Take provided measurement cup full of water (112ml) and soak one portion (pe-packed) of the powder for 12 hours, then boil it until the upper level has been reduced to 1/4, filter, cool down to room temperature, drink
  Interventions: Drug: Sida cordifolia roots; Drug: Phyllanthus niruri
- Modern extract herbal treatment (Experimental): Phyllanthus niruri extract 2 capsules 3 times a day with warm water before meals for 8 weeks
  Sida cordifolia roots extract 2 capsules 2 times a day with warm water before meals for 8 weeks
  Interventions: Drug: Sida cordifolia roots extract; Drug: Phyllanthus niruri extract
- Placebo (Placebo Comparator): Phyllanthus niruri placebo 2 capsules 3 times a day with warm water before meals for 3 weeks
  Sida cordifolia placebo 2 capsules 2 times a day with warm water before meals for 3 weeks
  Interventions: Other: Sida cordifolia placebo; Other: Phyllanthus niruri placebo

INTERVENTIONS:
Drug: Sida cordifolia roots — Sida cordifolia roots, crude drug (coarse powder) a plant product 7g (packages prepared) are soaked in 112ml water (measurement cup provided) for 12 hours and then boiled until the level is reduced to 1/4 of hight. Fluid is filtered an drunk after cooling down to room temperature - orally 2 times a day before breakfast and dinner
  Other Names: Bala moola; Bala
  Arms: Ancient herbal treatment
Drug: Phyllanthus niruri — Phyllanthus niruri (whole plant) fine powder 3g three times a day with warm water before meals taken orally.
  Other Names: Phyllanthus amarus; Bhumyamalaki; Tamalaki
  Arms: Ancient herbal treatment
Drug: Sida cordifolia roots extract — gelatine capsule with 300mg Sida cordifolia roots spraydry extract 12:1 concentrated normalized to alkaloids (alcoholic/aqueous extract) - 2 capsules taken orally 2 times a day with warm water before meal
  Other Names: Bala moola; Bala
  Arms: Modern extract herbal treatment
Drug: Phyllanthus niruri extract — gelatine capsule with 300mg Phyllanthus niruri spray dry extract 5:1 concentrated normalized to bitters (alcohol/aqueous extract) - 2 capsules taken orally 3 times a day with warm water before meal
  Other Names: Phyllanthus amarus; Bhumyamalaki; Tamalaki
  Arms: Modern extract herbal treatment
Other: Sida cordifolia placebo — 300mg inert Maltodextrin in gelatine capsule. 2 capsules given 2 times a day orally with warm water before meals
  Other Names: Placebo; Inert maltodextrine; Maltodextrine
  Arms: Placebo
Other: Phyllanthus niruri placebo — 300mg inert Maltodextrin in gelatine capsule. 2 capsules given 3 times a day orally with warm water before meals
  Other Names: Placebo; Inert Maltodextrin; Maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether phyllanthus niruri and sida cordifolia are effective in treatment of diabetic polyneuropathy compared to placebo. Also two different administration forms (extract capsules and crude herbs) are used to find out whether there are differences in efficiency and compliance.

DETAILED DESCRIPTION:
This study will explore the difference in therapeutic efficiency between modern extracts and whole drug powder of Phyllanthus niruri plus Sida cordifolia root decoction in diabetic neuropathy compared to placebo. The difference in compliance regarding medicine and food recommendations will be additionally documented.

Design - Study in two parts:

Part I: prospective, placebo-controlled, partly double-blinded (regarding 2 of the arms- all arms are investigator-blinded), 3 arm-parallel group study for 3 weeks Part II: prospective, investigator-blinded, long-term-study for 8 weeks. The active groups of part I will continue with their assigned medication and the placebo-patients of part I will be randomized again for the 2 groups of active medication.

Methods:

Symptoms will be assessed using Neuropathy total symptom score 6 (NTSS-6) as main primary parameter. Additional quantitative sensory testing will be done with the Neuropathy Analyzer Vibrotherm Dx from Diabetic Footcare India for detection of vibration and thermal sensation threshold. Tolerability, adverse drug reactions, Compliance regarding medication intake and dietary recommendations will be documented by an additional questionnaire.

Three randomized groups of 30 outpatients each (powder/decoction ; extract ; placebo) will be created for the part I of the study for the first 3 weeks.

At part I placebo group will be double blinded compared to extract group and investigator-blinded to powder/decoction group.

After 3 weeks the patients of the placebo group will be randomly assigned into both active treatment groups for part II to describe the course of treatment with both administration forms with 45 patients each.

Study visits will be prior and after 1,2,3,5 and 8 weeks.

Statistical plan: The primary parameter will be compared by Mann Whitney-U-Test.

Secondary Parameters will be descriptively analysed.

Implication:

A new herbal formulation will be tested for diabetic neuropathy with modern randomized placebo controlled study design in Part I. The outcome of the observation in part II will bring us closer to evidence based selection of different ayurvedic preparations in an upraising marked of new extraction technologies.

Registry procedures and other quality factors:

Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (medical records, paper case report forms).

Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.

Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* positive history of type 1 or 2 diabetes mellitus having the symptoms of diabetic neuropathy (sensory, peripheral) will be selected.
* Only outpatient setting will be included.
* Patients with ≥2 symptoms having at least one symptom with moderate severity in occasional frequency (3 points in NTSS-6) are included if they additionally show an impaired vibration detection threshold.

Exclusion Criteria:

* suffering from any other associated clinical conditions influencing peripheral nerve function, for example:
* peripheral vascular disease if reason for nerve damage
* vitamin deficiency (FOL,B12,E)
* heavy metal intoxication (especially with lead, cadmium and thallium)
* other intoxications (alcohol, medicine)
* infectious disease (like HIV, typhus, syphilis, lyme disease, mononucleosis,...)
* cancer
* autoimmune disease
* hepatitis
* vasculitis
* amyloidosis
* severe kidney failure
* pregnancy
* disorder of connective tissue
* steroids taken up to 1 month prior to study
* the likely need for insulin therapy

Regarding prior medication patients are advised not to start additional therapy during the study as long as symptoms are not worsening, antihyperglycaemic drugs will only be adjusted by study physicians if necessary.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Improvement of NTSS-6 SCORE in per cent from baseline | Initially, after 1, 2, 3, 5, 8 weeks of treatment, where placebo group will start again in one of the herbal treatment groups after 3 weeks (9 instead of 6 assessments)
  Validated symptom score containing 6 questions investigation severity (not present, mild, moderate, severe) and frequency (never or occasional, occasional but normal, often, almost continuous) of symptoms (aching pain, allodynia, burning pain, lancinating pain, numbness, prickling sensation).

SECONDARY OUTCOMES:
Improvement from baseline in per cent of quantitative sensory testing of vibration and thermal (hot/cold) threshold (score) | Initially, after 1, 2, 3, 5, 8 weeks of treatment, where placebo group will start again in one of the herbal treatment groups after 3 weeks (9 instead of 6 assessments)
  Semi-automated Neuropathy Analyser Dx from Diabetic Footcare India used to detect vibration and thermal (hot/cold) threshold (both soles)
  Inability to feel vibration up to: Normal: 10Hz below age of 50a and 15Hz above age of 50a = scoring "0"; Mild: 11-15Hz below age of 50a and 16-20Hz above age of 50a = scoring "1"; Moderate: 16-20Hz below age of 50a and 21-25Hz above age of 50a = scoring "2"; Severe: 20Hz below age of 50a and 26Hz above age of 50a = scoring "3"
  Inability to feel cold down to: Normal: 20°C = scoring "0"; Mild: 19-15°C = scoring "1"; Moderate: 14-10°C = scoring "2"; Severe: < 9°C = scoring "3"
  Inability to feel hot up to: Normal: 42°C = scoring "0"; Mild: 43-45°C = scoring "1"; Moderate: 46-48°C = scoring "2"; Severe: > 49°C = scoring "3"
  Temperature of the probe is to be reduced from 30°C to 0°C to record perception of cold sensation and temperature of the probe is to be increased from 30°C up to 50°C to record perception of heat sensations.
Assessment of compliance regarding medication and dietary recommendations (score). | After 1, 2, 3, 5, 8 weeks of treatment, where placebo group will start again in one of the herbal treatment groups after 3 weeks (8 instead of 5 assessments)
  The used questionaire is an adaption of the warfarin compliance-assessment scale from Community Anticoagulation Therapy Clinic in Iowa. (Huber, Levett, & Atkinson, 2008)
  Medication - Missed doses:
  No dose missed = score "0"
  One dose in a week missed = score "1"
  Two doses in a week missed = score "2"
  Three or more doses missed = score "3"
  Medication - Additional doses:
  No extra dose = score "0"
  One extra dose = score "1"
  Two extra doses = score "2"
  Three or more extra doses in a week = score "3"
  Food habits:
  Completely followed dietary recommendations = score "0"
  One day a week I ignored dietary recommendations = score "1"
  Two days a week I ignored dietary recommendations = score "2"
  Three or more days a week I ignored recommendations = score "3"

OTHER OUTCOMES:
Patient Diary | From start to end of treatment (8 weeks, 11 weeks for placebo group)
  With every distributed one-week-package of drug/placebo the patients will get a diary where they are supposed to fill in if medication has been taken (morning/lunch/dinner) and how there symptoms are like (non, mild, moderate, severe) for every single day.

CONTACTS AND LOCATIONS:
Overall Officials: Shivenarain N. Gupta, Prof. Dr., Principal Investigator — P.D. Patel Ayurveda Hospital / Rosenberg European Academy of Ayurveda
Locations (1):
- P.D. Patel Ayurveda Hospital, Nadiād, Gujarat, India

REFERENCES:
- [Background] Asare GA, Addo P, Bugyei K, Gyan B, Adjei S, Otu-Nyarko LS, Wiredu EK, Nyarko A. Acute toxicity studies of aqueous leaf extract of Phyllanthus niruri. Interdiscip Toxicol. 2011 Dec;4(4):206-10. doi: 10.2478/v10102-011-0031-9. PMID 22319255
- [Background] Bastyr EJ 3rd, Price KL, Bril V; MBBQ Study Group. Development and validity testing of the neuropathy total symptom score-6: questionnaire for the study of sensory symptoms of diabetic peripheral neuropathy. Clin Ther. 2005 Aug;27(8):1278-94. doi: 10.1016/j.clinthera.2005.08.002. PMID 16199253
- [Background] Boulton AJ. The diabetic foot: from art to science. The 18th Camillo Golgi lecture. Diabetologia. 2004 Aug;47(8):1343-53. doi: 10.1007/s00125-004-1463-y. Epub 2004 Jul 28. PMID 15309286
- [Background] Cornblath, DR. Diabetic neuropathy: Diagnostic methods. Advanced Studies in Medicine 4(8a):650-661, 2004.
- [Background] Dettori J. The random allocation process: two things you need to know. Evid Based Spine Care J. 2010 Dec;1(3):7-9. doi: 10.1055/s-0030-1267062. No abstract available. PMID 22956922
- [Background] Grover JK, Yadav S, Vats V. Medicinal plants of India with anti-diabetic potential. J Ethnopharmacol. 2002 Jun;81(1):81-100. doi: 10.1016/s0378-8741(02)00059-4. PMID 12020931
- [Background] Huber CS, Levett JM, Atkinson JM. A Tool to Assess Compliance in Anticoagulation Management. In: Henriksen K, Battles JB, Keyes MA, Grady ML, editors. Advances in Patient Safety: New Directions and Alternative Approaches (Vol. 3: Performance and Tools). Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK43677/ PMID 21249935
- [Background] Patel K, Patel M, Gupta SN. Effect of Atibalamula and Bhumyamalaki on thirty-three patients of diabetic neuropathy. Ayu. 2011 Jul;32(3):353-6. doi: 10.4103/0974-8520.93913. PMID 22529650
- [Background] Kanth VR, Diwan PV. Analgesic, antiinflammatory and hypoglycaemic activities of Sida cordifolia. Phytother Res. 1999 Feb;13(1):75-7. doi: 10.1002/(SICI)1099-1573(199902)13:13.0.CO;2-F. PMID 10189958
- [Background] Kastenbauer T, Sauseng S, Brath H, Abrahamian H, Irsigler K. The value of the Rydel-Seiffer tuning fork as a predictor of diabetic polyneuropathy compared with a neurothesiometer. Diabet Med. 2004 Jun;21(6):563-7. doi: 10.1111/j.1464-5491.2004.01205.x. PMID 15154940
- [Background] Konate K, Bassole IH, Hilou A, Aworet-Samseny RR, Souza A, Barro N, Dicko MH, Datte JY, M'Batchi B. Toxicity assessment and analgesic activity investigation of aqueous acetone extracts of Sida acuta Burn f . and Sida cordifolia L. (Malvaceae), medicinal plants of Burkina Faso. BMC Complement Altern Med. 2012 Aug 11;12:120. doi: 10.1186/1472-6882-12-120. PMID 22883637
- [Background] Kudom AA, Mensah BA, Botchey MA. Aqueous neem extract versus neem powder on Culex quinquefasciatus: implications for control in anthropogenic habitats. J Insect Sci. 2011;11:142. doi: 10.1673/031.011.14201. PMID 22233153
- [Background] Kumar P. S., et al. Immediate effects of nerve sliders and nerve massage on vibration and thermal perception thresholds in patients with painful diabetic peripheral neuropathy- a pilot randomized clinical trial. Physiotherapy and Occupational Therapy Journal 3(3):5-19, July - Sept 2010
- [Background] Sumanth M, Mustafa SS. Antistress, Adoptogenic Activity of Sida cordifolia Roots in Mice. Indian J Pharm Sci. 2009 May;71(3):323-4. doi: 10.4103/0250-474X.56027. PMID 20490305
- [Background] Neeraj, T., & Parul, S. (2011). Quality standards of indian medicinal plants. New Delhi: Indian Council of Medical Research, Medicinal Plants Unit.
- [Background] Shy ME, Frohman EM, So YT, Arezzo JC, Cornblath DR, Giuliani MJ, Kincaid JC, Ochoa JL, Parry GJ, Weimer LH; Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Quantitative sensory testing: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2003 Mar 25;60(6):898-904. doi: 10.1212/01.wnl.0000058546.16985.11. PMID 12654951
- [Background] Smieja M, Hunt DL, Edelman D, Etchells E, Cornuz J, Simel DL. Clinical examination for the detection of protective sensation in the feet of diabetic patients. International Cooperative Group for Clinical Examination Research. J Gen Intern Med. 1999 Jul;14(7):418-24. doi: 10.1046/j.1525-1497.1999.05208.x. PMID 10417599
- [Background] Srividya N, Periwal S. Diuretic, hypotensive and hypoglycaemic effect of Phyllanthus amarus. Indian J Exp Biol. 1995 Nov;33(11):861-4. PMID 8786163
- See also: Nadiad Ayurveda College and Hospital - Site of study — http://www.nadiadayurveda.org
- See also: Sponsor - Rosenberg European Academy of Ayurveda — http://www.ayurveda-akademie.org/en/home/
- See also: Funding society: European Professional Association of Ayurveda-Practitioners and -Therapists — http://www.ayurveda-verband.eu/?L=1